CLINICAL TRIAL: NCT06985004
Title: Predicting Operational Difficulties and Outcomes of Robot-Assisted Radical Prostatectomy (RARP) Based on Preoperative Assessment - Introducing the PIODO (Preoperative Index for Operative Difficulties and Outcomes) Questionnaire
Brief Title: Predicting Operational Difficulties and Outcomes of RARP Based on Preoperative Assessment - Introducing the PIODO Questionnaire
Status: Active, not recruiting | Type: Observational
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Sponsor
Other Study IDs: KB.006.121.2022/Z-110249
Record Dates: First submitted 2025-04-09; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer; Robot-Assisted Laparoscopic Radical Prostatectomy
Keywords: Prostate cancer; RARP; robot-assisted radical prostatectomy; preoperative assessment; pelvimetry; magnetic resonance imaging
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Consecutive patients with prostate cancer who underwent elective RARP
  Interventions: Other: PIODO Questionnaire

INTERVENTIONS:
Other: PIODO Questionnaire — An original PIODO Questionnaire is a structured protocol that has been developed by the investigators of this study for the preoperative assessment of patients undergoing RARP. It evaluates not only clinical data on the prostate cancer, but also patient characteristics, including anthropometric measurements of the pelvis. The aim is to develope a tool that can be used to predict the risk of operational difficulties and possible outcomes of RARP.

SUMMARY:
The goal of this observational study is to learn about the factors that affect the course of robot-assisted radical prostatectomy and have an impact on functional and oncological outcomes in patients undergoing RARP. The main question it aims to answer is:

• Can the investigators predict the occurrence of operational difficulties and outcomes of RARP based on preoperative assessment including body habitus and pelvimetry?

Participants undergoing RARP will be assessed preoperatively with the use of a PIODO Questionnaire, a structured protocol of preoperative assessment focusing on clinical data and MRI pelvic measurements to evaluate if the investigators can predict the risk of operational difficulties and possible outcomes of RARP. In a 1 year follow-up the investigators will collect data on functional and oncological outcomes.

DETAILED DESCRIPTION:
Various factors affect the course of RARP and have an impact on functional and oncological outcomes. To date, no structured protocol has been developed for the preoperative assessment of patients undergoing RARP that evaluates not only clinical data on the prostate cancer, but also patient characteristics, including anthropometric measurements of the pelvis. Based on our previous research and preliminary study, the investigators have developed a PIODO Questionnaire to assess these factors and verify whether it is possible to predict the occurrence of operative difficulties as well as functional and oncological outcomes.

Participants undergoing RARP will be assessed preoperatively using the PIODO Questionnaire. The investigators will collect medical data and pelvic MRI measurements to evaluate if the investigators can predict the risk of operational difficulties and possible outcomes of RARP. In a 1-year follow-up, the investigators will obtain information on potency and continence, as well as the presence of biochemical recurrence.

Achieving our goal will allow us to facilitate counselling of patients on their relative likelihood of post-operative continence or erectile function based on individual factors and anthropometric measurements and allow urologists to predict operative difficulties they may face during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with prostate cancer undergoing RARP.

Exclusion Criteria:

* Neoadjuvant androgen deprivation therapy before RARP.
* Lack of consent for study participation or willingness to comply with all procedures and assessments.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The investigators included in the study population consecutive patients with prostate cancer (diagnosis code C61 according to ICD-10 classification) who underwent elective RARP from January 2024 to December 2024 at the Department of Urology and Urological Oncology of Pomeranian Medical University in Szczecin.
Sampling Method: Non-Probability Sample
Enrollment: 288 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Preoperative Index for Operative Difficulties and Outcomes (PIODO Questionnaire) | Preoperatively
  Preoperative assessment of patients undergoing RARP using an original questionnaire. The sum of the points obtained is presented as a number. The minimum value is 10 and maximum value is 34. The investigators' assumption is that the higher the score, the more difficult the surgery and the worse the functional and oncological outcome.

SECONDARY OUTCOMES:
Angle between the pubic bone and the prostate | Preoperatively
  The angle between the pros¬tatic urethra and the posterior side of the pubic bone. Measured in degrees on MRI T2-weighted images.
Pubic symphysis-prostate apex length (PAL) | Preoperatively
  The distance between the extension lines of the suprapubic ridge line and the prostate apical line. Measured in centimeters on MRI T2-weighted images.
Membranous urethral length (MUL) | Preoperatively
  The upper limit of MUL is the lower border of the peripheral zone of the prostate, dorsal to the membranous urethra. The lower limit of MUL is the origin of the penile base at the dorsal side of the urethral lumen. Measured in milimeters on MRI T2-weighted images.
Protrusion of the prostate into the bladder | Preoperatively
  Evaluation of the presence or absence of protrusion of the prostate into the bladder. If the tip of the prostate protruded to the base of the urinary bladder, protrusion of the prostate into the bladder was considered present. Measured in milimeters on MRI T2-weighted images.
Anteroposterior diameter of the pelvic inlet (API) | Preoperatively
  Diameter from the sacral promontory to the most superior aspect of the pubic symphysis. Measured in centimeters on MRI T2-weighted images.
Pelvic depth (PD) | Preoperatively
  Diameter from the sacral promontory to the most inferior point of the pubic symphysis. Measured in centimeters on MRI T2-weighted images.
The anteroposterior distance at the midpelvis (APM) | Preoperatively
  Diameter from the inferior aspect of the pubic symphysis to the sacrococcygeal junction. Measured in centimeters on MRI T2-weighted images.
Pelvic outlet (APO) | Preoperatively
  Diameter from the inferior aspect of the pubic symphysis to the tip of the coccyx. Measured in centimeters on MRI T2-weighted images.
Anteroposterior diameter of the working space during surgery (Workspace AP) | Preoperatively
  Diameter from anterior peritoneum to anterior border of coccyx (inner border). Measured in centimeters on MRI T2-weighted images.
Transevrse diameter of the working space during surgery (Workspace T) | Preoperatively
  Diameter between medial border of acetabulum. Measured in centimeters on MRI T2-weighted images.

OTHER OUTCOMES:
Erectile function | Preoperatively and in 1 year follow-up after RARP.
  Measured with the use of International Index of Erectile Function-5 (IIEF-5). The minimum value is 0 and maximum value is 25. The higher the score the better erectile function.
Sexual activity | Preoperatively and in 1 year follow-up after RARP.
  Presence of sexual activity marked as 1, lack of sexual activity marked as 0.
Lower urinary tract symptoms (LUTS) | Preoperatively
  Presence of LUTS marked as 1, lack of symptoms marked as 0.
PSA | Preoperatively and in 1 year follow-up after RARP.
  Prostate-specific antigen (PSA) serum level.
Prostate volume | Preoperatively
  Prostate volume based on the MRI scan in milliliters.
Suspected prostate cancer on MRI | Preoperatively
  Measured using Prostate Imaging Reporting and Data System (PI-RADS) assessment categories.
Histopatology of prostate cancer | Preoperatively and up to 4 weeks after the surgery.
  Histological grading of adenocarcinoma of the prostate, including use of the International Society of Urological Pathology (ISUP) modified Gleason grades. The minimum value us 1 and maximum value is 5. The higher the score the more advanced cancer.
Clinical stage of prostate cancer | Preoperatively
  Stage based on digital rectal examination (DRE) only in accordance with the EAU guidelines.
Weight and height | Preoperatively
  Weight and height will be combined to report body mass index (BMI) in kg/m^2
Comorbidities | Preoperatively
  List of patients comorbidities.
Medications | Preoperatively
  Medications that can affect continence and/or erectile function - 1 if used, 0 if not.
Operative difficulties | Intraoperatively
  Operative difficulties were defined as:
  1. Operative time of 3 hours or longer.
  2. Blood loss over 500 ml.
  3. Need for blood transfusion during surgery.
  4. Lack of nerve-sparing unrelated to high-risk carcinoma.
  5. Presence of intraoperative complications reported by the surgeon. Presence of operative difficulties marked as 1, lack of difficulties as 0.
Postoperative complications | In 90 days follow-up after RARP.
  Precence of postoperative complications during first 90 days after RARP - 1 if occured, 0 if not.
Continence | In 1 year follow-up after RARP.
  Measured with the Urinary Domain of the Expanded Prostate Cancer Index Composite (EPIC). The minimum value is 6 and maximum value is 28. The higher score the worse continence.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology and Urological Oncology, Szczecin, Poland

IPD SHARING:
Plan to Share IPD: No